CLINICAL TRIAL: NCT03885544
Title: Effects of Consuming Red Meat on the Gut Microbiota in Young Adults
Acronym: S51
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 1709019738
Record Dates: First submitted 2018-03-27; First posted 2019-03-21 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-07

CONDITIONS: Diet Modification
Keywords: beef; pork; red meat; gut microbiota

STUDY DESIGN:
Intervention Model Description: This is a 24-week randomized controlled, crossover, single-blind study. Following a 5-wk pre-intervention baseline period, subjects will be randomly assigned to consume a controlled diet that either does not contain any red meat (lacto-ovo vegetarian, LOV), or contains unprocessed lean red meat, or contains processed lean red meat, for 3 weeks. After a 5-week dietary 'washout' period, they will consume one of the alternative diets for 3 weeks. After the second 5-week dietary 'washout' period, they will consume the remaining alternative diet for 3 weeks. Stool and fasting-state blood samples will be obtained at the end of study weeks 3, 4, 7, 8, 11, 12, 15, 16, 19, 20, 23, and 24, which correspond to before and during the last 2 weeks of the three 3-wk controlled diet periods. Consecutive 4-day 24-hour urine samples will be collected within the assessment weeks of each dietary 'washout' period and control diet period (study weeks 4, 8, 12, 16, 20, 24).
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Controlled lacto-ovo vegetarian diet (Active Comparator): Subjects will be randomized and assigned into an intervention to consume the controlled lacto-ovo vegetarian diet without red meat for 3 weeks.
  Interventions: Other: Controlled Lacto-ovo vegetarian diet
- Controlled unprocessed red meat diet (Experimental): Subjects will be randomized and assigned into an intervention to consume the controlled lacto-ovo vegetarian diet with unprocessed red meat for 3 weeks.
  Interventions: Other: Controlled Unprocessed red meat diet
- Controlled processed red meat diet (Experimental): Subjects will be randomized and assigned into an intervention to consume the controlled lacto-ovo vegetarian diet with processed red meat for 3 weeks.
  Interventions: Other: Controlled processed red meat diet

INTERVENTIONS:
Other: Controlled Lacto-ovo vegetarian diet — Subjects will be randomized and assigned into an intervention to consume the controlled lacto-ovo vegetarian (LOV) diet for 3 weeks. All foods will be provided to subjects during the intervention. Each subject's energy requirement will be estimated using sex-specific equations published by the Institute of Medicine for weight maintenance during the intervention.
  Arms: Controlled lacto-ovo vegetarian diet
Other: Controlled Unprocessed red meat diet — The unprocessed red meat diet will be the same as the LOV diet except that one 3-ounce portion of unprocessed red meat per day, 7 days per week (21 oz/wk) will be included. The unprocessed red meat will include beef tenderloin and pork loin. All foods will be provided to subjects during the intervention.
  Arms: Controlled unprocessed red meat diet
Other: Controlled processed red meat diet — The processed red meat diet will be the same as the LOV diet except that one 3-ounce portion of processed red meat per day, 7 days per week (21 oz/wk) will be included. The processed red meat will include a variety of beef and pork luncheon meats with different methods of preservation. All foods will be provided to subjects during the intervention.
  Arms: Controlled processed red meat diet

SUMMARY:
The purpose of this study is to assess the impact of consuming unprocessed and processed red meat on gut microbiota in young healthy adults in a cross-over, randomized controlled feeding trial.

DETAILED DESCRIPTION:
The purpose of this study is to assess the impact of consuming processed and unprocessed red meat on gut microbiota in young healthy adults in a cross-over, randomized controlled feeding trial. The hypothesis is that compared to consuming a meat-free lacto-ovo vegetarian (LOV) diet, (1) consuming the LOV diet with unprocessed red meat or processed red meat (omnivorous diet) will shift the gut microbiota with greater abundance of the bacteria Lactobacillus and other SCFA producers such as Clostridium XIVa, and no increase of pathogenic bacteria. The concentration of SCFA in stools will also increase in subjects consuming the unprocessed red meat diet. Compared to consuming a meat-free lacto-ovo vegetarian (LOV) diet, (2) consuming the LOV diet with processed beef and pork (omnivorous diet) will result in a comparable shift in gut microbiota as unprocessed red meat, except for greater abundance of taxa Erysipelotrichaceae and lower abundance of Lachnospiraceae.

ELIGIBILITY:
Inclusion Criteria:

* male or female,
* 20-35 years old,
* BMI 20.0-29.9 kg/m2,
* fasting serum total cholesterol <240 mg/dL, low-density lipoprotein cholesterol <160 mg/dL, triglycerides <400 mg/dL, and glucose <110 mg/dL;
* systolic/diastolic blood pressure <140/90 mmHg;
* body weight stable for 3 months prior (±3 kg); stable physical activity regimen 3 months prior;
* medication use stable for 6 months prior and not using medications or supplements known to impact gut function;
* on-smoking; not drinking more than 2 alcoholic drinks per day;
* non-diabetic,
* no history of gastrointestinal disorders, surgeries or cancers;
* non-pregnant and not lactating.
* Participants must be willing and able to consume the prescribed diets (lacto-ovo vegetarian and omnivorous).

Exclusion Criteria:

* male or female < 20->35 years old,
* BMI <20.0- >29.9 kg/m2,
* fasting serum total cholesterol >240 mg/dL, low-density lipoprotein cholesterol >160 mg/dL, triglycerides >400 mg/dL, and glucose >110 mg/dL;
* systolic/diastolic blood pressure >140/90 mmHg;
* body weight stable for <3 months prior (±3 kg);
* stable physical activity regimen < 3 months prior;
* medication use unstable for 6 months prior and using medications or supplements known to impact gut function;
* smoking;
* drinking more than 2 alcoholic drinks per day;
* diabetic,
* history of gastrointestinal disorders, GI surgeries or GI cancers;
* pregnant or lactating.

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2018-01-09 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Changes in gut microbiota composition | 21 months. Stool samples will be obtained at the end of study weeks 3, 4, 7, 8, 11, 12, 15, 16, 19, 20, 23, and 24, which correspond to before and during the last 2 weeks of the three 3-wk controlled diet periods.
  The hypothesis is that compared to consuming a meat-free lacto-ovo vegetarian (LOV) diet, (1) consuming the LOV diet with unprocessed red meat or processed red meat (omnivorous diet) will shift the gut microbiota with greater abundance of the bacteria Lactobacillus and other SCFA producers such as Clostridium XIVa, and no increase of pathogenic bacteria. Compared to consuming a meat-free lacto-ovo vegetarian (LOV) diet, (2) consuming the LOV diet with processed beef and pork (omnivorous diet) will result in a comparable shift in gut microbiota as unprocessed red meat, except for greater abundance of taxa Erysipelotrichaceae and lower abundance of Lachnospiraceae.
Concentrations of short chain fatty acids (SCFA) | 21 months. Stool samples will be obtained at the end of study weeks 3, 4, 7, 8, 11, 12, 15, 16, 19, 20, 23, and 24, which correspond to before and during the last 2 weeks of the three 3-wk controlled diet periods.
  The hypothesis is that compared to consuming a meat-free lacto-ovo vegetarian (LOV) diet, the concentration of SCFA in stools will also increase in subjects consuming the unprocessed or processed red meat diet.

OTHER OUTCOMES:
metabolomics analysis | Undecided.
  Saves of blood, urine, and stool samples will be kept for possible further metabolomics and foodomics analyses.

CONTACTS AND LOCATIONS:
Overall Officials: Wayne W Campbell, Ph.D., Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

REFERENCES:
- [Derived] Wang Y, Lindemann SR, Cross TL, Tang M, Clark CM, Campbell WW. Effects of Adding Lean Red Meat to a U.S.-Style Healthy Vegetarian Dietary Pattern on Gut Microbiota and Cardiovascular Risk Factors in Young Adults: a Crossover Randomized Controlled Trial. J Nutr. 2023 May;153(5):1439-1452. doi: 10.1016/j.tjnut.2023.03.013. Epub 2023 Mar 14. PMID 36921804